CLINICAL TRIAL: NCT07401420
Title: Project Plan Physicians' Experiences of the Decision-making Process Regarding Decisions to Withhold/Discontinue Life-sustaining Treatment in Children Cared for in Intensive Care Units in Sweden. A Qualitative Study.
Brief Title: Life Sustaining Treatments in Critically Ill Children
Acronym: LST-Ped-Int
Status: Not yet recruiting | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: LST-Ped-Int
Record Dates: First submitted 2026-01-19; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Critical Illness; Ethics; End of Life Care
Keywords: Critical illness; Ethics; End of life care
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intensive care physicians: Intensive care physicians
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — Observational study

SUMMARY:
Summary of the Research on Withdrawing and Withholding Life-Sustaining Treatment for Critically Ill Children Background Medical treatments require regular evaluation to ensure they align with the patient's best interests, particularly in intensive care where quality of life is often compromised. In the context of critically ill children, the challenge increases as patients may not be fully conscious or capable of expressing their needs and preferences. While intensive care can extend life, end-of-life situations necessitate careful consideration to avoid providing futile treatments that do not benefit the patient.

Decision-Making Complexity Identifying when further treatment is beneficial poses significant challenges, influenced by various factors including the wishes of the patient and guardians. Previous studies indicate variability among healthcare providers in treatment decisions, often stemming from personal experiences and emotional responses. However, comparable research focusing on critically ill children in Nordic contexts remains scarce. Medical decisions often require balancing potential benefits against the risks of extended suffering or loss of valuable time at the end of life.

A previous survey on end-of-life care in Europe indicated similar attitudes across regions but highlighted the need for cultural considerations. Sweden's distinct social and cultural values, characterized by individualism and secularism, may influence practices surrounding life-sustaining treatment.

Research Aims This research aims to investigate the factors affecting decision-making regarding the withdrawal and withholding of life-sustaining treatments for critically ill children in Swedish and Nordic intensive care units (ICUs). It will examine practitioners' experiences, attitudes, and the relative impact of children's autonomy in these decisions, excluding neonatal care.

Key scientific questions focus on Physicians' attitudes and challenges regarding treatment withdrawal.

Methodology

Semi-structured interviews in multiple ICUs to explore ethical dilemmas faced by physicians.

DETAILED DESCRIPTION:
Summary of the Research on Withdrawing and Withholding Life-Sustaining Treatment for Critically Ill Children Background Medical treatments require regular evaluation to ensure they align with the patient's best interests, particularly in intensive care where quality of life is often compromised. In the context of critically ill children, the challenge increases as patients may not be fully conscious or capable of expressing their needs and preferences. While intensive care can extend life, end-of-life situations necessitate careful consideration to avoid providing futile treatments that do not benefit the patient.

Decision-Making Complexity Identifying when further treatment is beneficial poses significant challenges, influenced by various factors including the wishes of the patient and guardians. Previous studies indicate variability among healthcare providers in treatment decisions, often stemming from personal experiences and emotional responses. However, comparable research focusing on critically ill children in Nordic contexts remains scarce. Medical decisions often require balancing potential benefits against the risks of extended suffering or loss of valuable time at the end of life.

A previous survey on end-of-life care in Europe indicated similar attitudes across regions but highlighted the need for cultural considerations. Sweden's distinct social and cultural values, characterized by individualism and secularism, may influence practices surrounding life-sustaining treatment.

Research Aims This research aims to investigate the factors affecting decision-making regarding the withdrawal and withholding of life-sustaining treatments for critically ill children in Swedish and Nordic intensive care units (ICUs). It will examine practitioners' experiences, attitudes, and the relative impact of children's autonomy in these decisions, excluding neonatal care.

Key scientific questions focus on Physicians' attitudes and challenges regarding treatment withdrawal.

Methodology

Semi-structured interviews in multiple ICUs to explore ethical dilemmas faced by physicians.The research question will be investigated through semi-structured individual interviews with physicians who work with children in intensive care units. This will include both intensive care specialists and physicians from other specialties, primarily pediatricians. Recruitment will involve contacting the four children's departments in Sweden to seek voluntary study participants. The children's clinics at the same hospitals will also be contacted to reach out to potential volunteers. Recruitment will thereafter proceed through repeated contact and snowballing, where interviewed participants will assist in the recruitment process.An interview guide will be created and piloted with three people for validation. Subsequently, the interview guide will be updated.

The interviews will be conducted via links and verbatim transcription with the help of speech recognition software, which will be connected to the interviewer during the interview. Analysis will occur in NVivo using Qualitative Content Analysis according to Granheim and Lundman, based on narrative theory.

ELIGIBILITY:
Inclusion Criteria:

* Specialist physicians in critical care with experience from end of life care in critically ill children.

Exclusion Criteria:

None

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Specialist physicians in critical care with experience from end of life care in critically ill children.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Physicians' attitudes and challenges regarding treatment withdrawal. | Interviews will be about 60 minutes
  Observational qualitative study with semi-structured interviewsanalysed with thematic analyses

IPD SHARING:
Plan to Share IPD: Yes
All IPD that cannot be traced to an individual person.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon reasonable request
Access Criteria: Upon reasonable request
URL: http://Datawillnotbesharedonawebsite

REFERENCES:
- [Background] Malhotra AK, Shakil H, Smith CW, Sader N, Ladha K, Wijeysundera DN, Singhal A, Kulkarni AV, Wilson JR, Witiw CD, Nathens AB. Withdrawal of Life-Sustaining Treatment for Pediatric Patients With Severe Traumatic Brain Injury. JAMA Surg. 2024 Mar 1;159(3):287-296. doi: 10.1001/jamasurg.2023.6531. PMID 38117514
- [Background] Zhong Y, Cavolo A, Labarque V, Gastmans C. Physicians' attitudes and experiences about withholding/withdrawing life-sustaining treatments in pediatrics: a systematic review of quantitative evidence. BMC Palliat Care. 2023 Sep 29;22(1):145. doi: 10.1186/s12904-023-01260-y. PMID 37773128
- [Background] Zhong Y, Cavolo A, Labarque V, Gastmans C. Physician decision-making process about withholding/withdrawing life-sustaining treatments in paediatric patients: a systematic review of qualitative evidence. BMC Palliat Care. 2022 Jun 24;21(1):113. doi: 10.1186/s12904-022-01003-5. PMID 35751075
- See also: Related Info — https://portal.icuregswe.org/utdata/2013-2023

DOCUMENTS (1):
  • Study Protocol (2026-01-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT07401420/Prot_000.pdf